CLINICAL TRIAL: NCT04099784
Title: Follow-up of Children Born From Freeze-only Versus Fresh Embryo Transfer: a Follow-up of a Randomized Controlled Trial
Brief Title: Health of Frozen Transferred Versus Fresh Transferred Children
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CS/BVMĐ/19/08
Record Dates: First submitted 2019-09-14; First posted 2019-09-23 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2019-11

CONDITIONS: Infertility; IVF
Keywords: Fresh transfer, freeze-only, ASQ-3, health of children
MeSH Terms: conditions — Infertility | interventions — Health Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Freeze-only: Children born from freeze-only group and frozen embryo transfer
  Interventions: Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Other: Developmental Red flags
- Fresh: Children born from fresh embryo transfer
  Interventions: Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Other: Developmental Red flags

INTERVENTIONS:
Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3 — Ages & Stages Questionnaires®, Third Edition (ASQ®-3) is a developmental screening tool designed for use by early educators and health care professionals. It relies on parents as experts, is easy-to-use, family-friendly and creates the snapshot needed to catch delays and celebrate milestones.
Other: Physical development and General Health — Physical development and General health examination
Other: Developmental Red flags — Developmental Red flags Questionnaires

SUMMARY:
In order to give strong recommendation on the efficacy and safety of fresh versus frozen embryo transfer, we conduct this study in order to investigate the physical and mental development of children from fresh versus frozen embryo transfer. Based on our Freeze-only study (Vuong et al., 2018), the women without polycystic ovary syndrome undergoing the first or second IVF were randomly assigned to receive either fresh or frozen embryos on day 3 after oocyte retrieval, which leads to the similarity in characteristics of these two groups. Hence, the result from analysing these offsprings would be preciously valuable.

DETAILED DESCRIPTION:
Since the first live birth after the transfer of a frozen-thawed embryo reported in 1984, cryopreservation has been considered as an enormous revolution in assisted reproductive technology (ART). It is observed that the trend of ART cycles using frozen embryo transfer is on the increase, which leads to a great deal number of children born from frozen embryos. This is the commencement of 2 embryo transfer strategies, the first one is transferring the fresh embryos, the other is freezing all the embryos and transfer them in the next cycle.

Comparing these two strategies, up till now, there are 4 published randomized control trials (RCTs) indicating different methods for certain groups of patients (Chen et al., 2016; Shi et al., 2018; Vuong et al., 2018; Wei et al., 2019). Regarding the efficacy, the freeze-all strategy outweighs the fresh embryo transfer in women with polycystic ovary syndrome (PCOS). While that efficacy gets a controversy in non-PCOS or ovulatory patients; two groups of authors indicated that these 2 strategies are equally effective, while the other group claims that the better result goes to cycles with frozen embryos. In term of safety, the rate of ovarian hyperstimulation syndrome (OHSS) is the equivalent or lower in the freeze-all group, which implies the important role of embryo-freezing in avoiding maternal risk. The question that whether freezing the embryos exerts effect on offspring is not thoroughly understood. The mostly used parameter in evaluating the safety of children is the perinatal status of infants, not the development of these children.

Searching literature, in 2010, S. Pelkonen published a large cohort study indicating that freezing the embryos do not change the rate of prematurity, low birthweight and being small for gestational age (Pelkonen et al., 2010). Looking further in our freeze-only study, our sub-analysis indicates that the livebirth weight of infants born from frozen embryos is 300 gram heavier than that from fresh embryos (Vuong et al., 2018). Following 4 studies comparing fresh and frozen embryo transfer, children from frozen embryos are similar or higher in term of newborn weight, and there is no study investigate the onward development of childrens born from these two strategies. The only proof on the development of children born from fresh verus frozen embryo is from one study with no randomization which states that children from fresh and frozen embryos share similar academic performance at the age 15-16 (Spangmose et al., 2019). We found no study investigate the impact of different embryo transfer strategies on the growth of children resulting from either fresh or frozen embryos.

In order to give strong recommendation on the efficacy and safety of fresh versus frozen embryo transfer, we conduct this study in order to investigate the physical and mental development of children from fresh versus frozen embryo transfer. Based on our Freeze-only study (Vuong et al., 2018), the women without polycystic ovary syndrome undergoing the first or second IVF were randomly assigned to receive either fresh or frozen embryos on day 3 after oocyte retrieval, which leads to the similarity in characteristics of these two groups. Hence, the result from analysing these offsprings would be preciously valuable.

ELIGIBILITY:
Inclusion Criteria:

* Live babies born from the first transfer of both freeze-only and fresh embryo transfer group from our Freeze-only study.
* Parents agree to participate in the study.

Exclusion Criteria:

* Babies died after perinatal period.

Ages: 1 Month to 66 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Live babies born following the frozen embryo transfer and fresh embryo transfer from our Freeze-only study (NCT02471573)
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
The average total ASQ-3 score | Up to 66 months after birth
  ASQ-3 (Ages and Stages Questionaires®) has 5 aspects: Communication, Gross motor, Fine motor, Problem solving and Personal-Social Each aspect has 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  ASQ-3 average = average score of 5 aspects.

SECONDARY OUTCOMES:
Score of Communication | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Gross motor | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
Score of Fine motor | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
Score of Problem solving | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
Score of Personal-Social | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
The rate of children who have at least one red flag sign | From 2 to 5.5 years after birth
  He or she has at least one red flag sign by age
  From 2 to < 3 year-old:
  * Has very unclear speech
  * Doesn't understand simple instruction • Doesn't speak in sentences
  * Doesn't make eye contact
  * Loses skills he/she once had
  From 3 to < 4 year-old:
  * Can't jump in place
  * Doesn't play pretend or make-believe • Speaks unclearly
  * Can't retell a favorite story
  * Doesn't use "me" and "you" correctly
  * Loses skills he/she once had
  From 4 to < 5.5 year-old:
  * Is easily distracted, has trouble focusing on one activity for more than 5 minutes • Doesn't talk about daily activities or experiences
  * Shows extreme behavior
  * Loses skills he/she once had
Duration of breast-feeding | Up to 24 months after birth
  Duration of breast-feeding
Infant age at which weaning starts | Up to 24 months after birth
  Infant age at which weaning starts
Name of diseases that lead to hospital admission | Up to 66 months after birth
  Name of diseases that lead to hospital admission
Number of hospital admission | Up to 66 months after birth
  Number of hospital admission
Weight | Through study completion, an average of 1.5 months
  Weight on the examination date
Height | Through study completion, an average of 1.5 months
  Height on the examination date

OTHER OUTCOMES:
Gestational age at delivery | At birth
  Gestational age at delivery
Mode of delivery | At birth
  Vaginal birth or C-section
Birth weight | At birth
  Weight of baby born
Length circumference | At birth
  Head circumference after birth Head circumference after birth Head circumference after birth Length circumference after birth
Head circumference | At birth
  Head circumference after birth
Rate of congenital anomalies | At birth
  Any congenital anomalies detected in baby born
Length of neonatal intensive care unit (NICU) admission | Up to 28 days after birth
  Number of admission days to NICU
Rate of Respiratory distress syndrome | Up to 28 days after birth
  Respiratory distress syndrome (RDS), diagnosed as the presence of tachypnoea >60/minute, sternal recession and expiratory grunting, need for supplemental oxygen, and a radiological picture of diffuse reticulogranular shadowing with an air bronchogram
Rate of Periventricular haemorrhage | Up to 28 days after birth
  Periventricular haemorrhage II B or worse, will be diagnosed by repeated neonatal cranial ultrasound by the neonatologist according to the guidelines on neuro-imaging described by de Vries et al.
Rate of Necrotizing enterocolitis | Up to 28 days after birth
  Necrotizing enterocolitis (NEC) will be diagnosed according to Bell.
Rate of Proven sepsis | Up to 28 days after birth
  Proven sepsis, will be diagnosed on the combination of clinical signs and positive blood cultures.
Rate of Composite of poor perinatal outcomes | Up to 28 days after birth
  Composite of poor perinatal outcomes, defined as intraventricular haemorrhage, respiratory distress syndrome, necrotizing enterocolitis or neonatal sepsis.
The rate of long-term illness and chronic conditions | Up to 66 months after birth
  Any long-term illness and chronic condition appears in a child

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Tan Binh, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen ZJ, Shi Y, Sun Y, Zhang B, Liang X, Cao Y, Yang J, Liu J, Wei D, Weng N, Tian L, Hao C, Yang D, Zhou F, Shi J, Xu Y, Li J, Yan J, Qin Y, Zhao H, Zhang H, Legro RS. Fresh versus Frozen Embryos for Infertility in the Polycystic Ovary Syndrome. N Engl J Med. 2016 Aug 11;375(6):523-33. doi: 10.1056/NEJMoa1513873. PMID 27509101
- [Background] Shi Y, Sun Y, Hao C, Zhang H, Wei D, Zhang Y, Zhu Y, Deng X, Qi X, Li H, Ma X, Ren H, Wang Y, Zhang D, Wang B, Liu F, Wu Q, Wang Z, Bai H, Li Y, Zhou Y, Sun M, Liu H, Li J, Zhang L, Chen X, Zhang S, Sun X, Legro RS, Chen ZJ. Transfer of Fresh versus Frozen Embryos in Ovulatory Women. N Engl J Med. 2018 Jan 11;378(2):126-136. doi: 10.1056/NEJMoa1705334. PMID 29320646
- [Background] Vuong LN, Dang VQ, Ho TM, Huynh BG, Ha DT, Pham TD, Nguyen LK, Norman RJ, Mol BW. IVF Transfer of Fresh or Frozen Embryos in Women without Polycystic Ovaries. N Engl J Med. 2018 Jan 11;378(2):137-147. doi: 10.1056/NEJMoa1703768. PMID 29320655
- [Background] Wei D, Liu JY, Sun Y, Shi Y, Zhang B, Liu JQ, Tan J, Liang X, Cao Y, Wang Z, Qin Y, Zhao H, Zhou Y, Ren H, Hao G, Ling X, Zhao J, Zhang Y, Qi X, Zhang L, Deng X, Chen X, Zhu Y, Wang X, Tian LF, Lv Q, Ma X, Zhang H, Legro RS, Chen ZJ. Frozen versus fresh single blastocyst transfer in ovulatory women: a multicentre, randomised controlled trial. Lancet. 2019 Mar 30;393(10178):1310-1318. doi: 10.1016/S0140-6736(18)32843-5. Epub 2019 Feb 28. PMID 30827784
- [Background] Pelkonen S, Koivunen R, Gissler M, Nuojua-Huttunen S, Suikkari AM, Hyden-Granskog C, Martikainen H, Tiitinen A, Hartikainen AL. Perinatal outcome of children born after frozen and fresh embryo transfer: the Finnish cohort study 1995-2006. Hum Reprod. 2010 Apr;25(4):914-23. doi: 10.1093/humrep/dep477. Epub 2010 Feb 2. PMID 20124395
- [Background] Spangmose AL, Malchau SS, Henningsen AA, Forman JL, Rasmussen S, Loft A, Schmidt L, Pinborg A. Academic performance in adolescents aged 15-16 years born after frozen embryo transfer compared with fresh embryo transfer: a nationwide registry-based cohort study. BJOG. 2019 Jan;126(2):261-269. doi: 10.1111/1471-0528.15484. Epub 2018 Oct 24. PMID 30276983
- [Derived] Vuong LN, Ly TT, Nguyen NA, Nguyen LMT, Le XTH, Le TK, Le KTQ, Le TV, Nguyen MHN, Dang VQ, Norman RJ, Mol BW, Ho TM. Development of children born from freeze-only versus fresh embryo transfer: follow-up of a randomized controlled trial. Fertil Steril. 2020 Sep;114(3):558-566. doi: 10.1016/j.fertnstert.2020.04.041. Epub 2020 Jun 16. PMID 32560970